CLINICAL TRIAL: NCT02761499
Title: Prospective Post Approval Clinical Follow-Up Study of the Commercially Available U-Motion II+ Acetabular System and UTF Reduced Stem
Brief Title: Post Approval Study of the Commercially Available U-Motion II+ Acetabular System and UTF Reduced Stem
Acronym: U-Move
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: United Orthopedic Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-2015
Record Dates: First submitted 2016-04-15; First posted 2016-05-04 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Hip Arthroplasty: The United Hip System consist of several components, and for this clinical evaluation it includes the U-Motion II+ Acetabular System (1) U-Motion II+ acetabular cup, (2) U-Motion II+ acetabular liner, (3) Cobalt-Chrome or BIOLOX delta ceramic femoral heads, and the 4) UTF Reduced Stem.
  Interventions: Device: U-Motion II+ Acetabular System

INTERVENTIONS:
Device: U-Motion II+ Acetabular System — U-Motion II+ Acetabular System (1) U-Motion II+ acetabular cup, (2) U-Motion II+ acetabular liner, (3) Cobalt-Chrome or BIOLOX delta ceramic femoral heads, and the 4) UTF Reduced Stem

SUMMARY:
This is a prospective, single arm, multi-center, post-approval study designed to evaluate the short and long term clinical performance and safety in subjects receiving primary total hip arthroplasty (THA) with the U-Motion II+ Acetabular System and UTF Reduced Stem.

DETAILED DESCRIPTION:
This is a prospective, single arm, multi-center, post-approval study designed to evaluate the short and long term clinical performance and safety in subjects receiving primary total hip arthroplasty (THA) with the U-Motion II+ Acetabular System and UTF Reduced Stem. The acetabular and femoral components will be uncemented. Study outcomes will be analyzed and published when 1.) all enrolled and implanted subjects complete their 6-week follow up, 2.) all implanted subjects complete their 2-year follow up, 3.) at the conclusion of the study.

It is anticipated that up to 200 subjects will be enrolled at up to 5 sites. The subjects will be evaluated at predetermined intervals: baseline, procedure/ discharge and 6 weeks, 3 months, 6 months, 12 months, and 24 months post treatment for primary analysis and annually up to 5 years for device survivorship. The estimated study duration from first enrollment through completion of the final report is expected to be approximately 7 years.

This study will be conducted at up to 5 investigational sites in the United States with previous clinical research experience and with adequate population of orthopedic patients requiring primary total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be considered for inclusion in the study.

1. Subject is between 18 and 75 years of age
2. Subject is indicated for a unilateral or bilateral total hip arthroplasty (THA) based on the approved labeling of the device
3. Subject has no history of previous prosthetic replacement device or orthopedic surgeries on the operative hip
4. Subject is willing and able to provide informed consent to participate in the study;
5. Subject is willing and able to understand the purpose of the study, his/her role, and is available to return to the clinic/hospital for all required follow-up visits;

Exclusion Criteria:

* Subjects will be excluded if, in the opinion of the Investigator, the subject does not qualify based on approved labeling requirements or Subject Inclusion criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects presenting with a documented history with chronic hip pain and disability due to degenerative joint disease such as osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2023-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Operative Success | 2 Years
  Post-operative increase in Harris Hip Score of > 20 points + radiographically stable implant + no additional femoral reconstruction stable implant + no additional femoral reconstruction

SECONDARY OUTCOMES:
Operative Time | Procedure
  Operative time in minutes
VAS Hip Pain | Baseline, Procedure, 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  Improvement in Hip Pain VAS scores out to 5 years
Device Related Adverse Events | Procedure, 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  Device related adverse events will be assessed at each follow up visit.
Length of hospital stay | 2 Years
  Length of stay in hours or days
Estimated Blood Loss (EBL) | 2 Years
  Estimated blood loss in cc's
HOOS Questionnaire | Baseline, Procedure, 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  To assess patient-relevant outcomes in five separate subscales (pain, symptoms, activity of daily living, sport and recreation function and hip related quality of life).
Subject Satisfaction | Procedure, 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  To assess the subject's satisfaction with their hip implant
Harris Hip Score | Baseline, Procedure, 6 weeks, 3 months, 6 months, 12 months, 2 Years, 3 Years, 4 Years and 5 Years.
  Assess outcome of total hip replacement

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Su, MD, Principal Investigator — HSS
Locations (6):
- United States (6):
  - Jacksonville Orthopaedic Institute, Jacksonville, Florida
  - Joint Replacement Institute, Naples, Florida
  - Hospital for Special Surgery, New York, New York
  - Ortho Dayton, Dayton, Ohio
  - Penn Orthopaedics, Philadelphia, Pennsylvania
  - Kenosha Orthopedics, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided